CLINICAL TRIAL: NCT01734369
Title: Environmental Risk Factors for the Development of Myositis in Military Personnel
Brief Title: Environmental Risk Factors for Myositis in Military Personnel
Status: Completed | Type: Observational
Sponsor: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 130015; 13-E-0015
Record Dates: First submitted 2012-11-22; First posted 2012-11-27 (Estimated); Last update posted 2025-12-31 (Actual); Status verified 2025-03-20

CONDITIONS: Dermatomyositis; Adult Polymyositis; Inclusion Body Myositis; Myositis
Keywords: Dermatomyositis; Inclusion Body Myositis; Myositis; Polymyositis; Military; Natural History
MeSH Terms: conditions — Dermatomyositis; Polymyositis; Myositis, Inclusion Body; Myositis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy Control Subjects: Military service members active duty or no longer in duty, military contractors, and civilians working for the military. Controls should be without a recognized autoimmune or chronic muscle disease.
- Myositis Subjects: Diagnosis of myositis during military service or service as a military contractor or civilian working for the military with polymyositis, dermatomyositis, or inclusion body myositis.

SUMMARY:
Background:

* Myositis is a rare disease in which the body s immune cells attack the muscle tissue. It can cause muscle weakness, swelling, and pain. It can develop in people with no history of muscle problems. Environmental exposures may determine who develops myositis. Genes may also affect development of the disease.
* Some people who serve in the military develop myositis. However, other military personnel do not. Researchers want to compare military personnel with and without myositis. They will look for common factors that might have led to the disease.

Objectives:

- To study environmental risk factors for myositis in military personnel.

Eligibility:

* Military personnel who developed myositis during their period of service.
* Healthy military personnel who do not have myositis or another autoimmune disease.

Design:

* Participants will have a physical exam and medical history.
* Participants will fill out forms about environmental exposures, particularly while in the military. The questions will ask about past infections, vaccines and medications, and personal habits. They will also ask about participants occupations during military service and their deployments.
* Participants will also provide blood samples for study.
* No treatment will be provided as part of this study.

DETAILED DESCRIPTION:
Myositis, an autoimmune muscle disease, likely develops as a result of environmental exposures in genetically susceptible persons. Preliminary data suggest a trend for an increasing incidence in myositis in military personnel over the last decade for unknown reasons. Although a few environmental exposures have been preliminarily associated with myositis in the civilian population, these have not been confirmed. In addition, no study has assessed exposures that might result in the development of myositis in military personnel. Military personnel experience a number of intense, unique exposures, often over a relatively short interval, which include different stresses, novel vaccines, distinct occupational exposures, battlefield injuries and unique chemicals during field deployment, that differ from those exposures in non-military populations. Therefore, we propose a protocol that consists of three complementary approaches to attempt to determine the environmental factors associated with the development of myositis in active duty military personnel and an initial understanding of the possible mechanisms involved. In the first approach, we will assess risk factors in a case-control study of 300 patients who developed myositis while on active duty by comparing them to 1500 active duty military personnel (randomly selected, but matched 5:1 by gender, race, and age and military service within 10 years) who have not been diagnosed with an autoimmune disease or chronic muscle disease. For this first approach, we will analyze existing military databases for information on medications, vaccines, infections, co-existing medical conditions, military occupations, deployments, and worldwide active duty locations. In the second case-control approach, we will attempt to define environmental factors associated with the development of myositis that developed in military personnel (n=150) by comparing them to 150 similarly matched military personnel who have not been diagnosed with an autoimmune disease or chronic muscle disease. This second approach will differ from the first approach, in that subjects will be prospectively enrolled and assessed during a single clinic visit to confirm diagnoses and examine patient questionnaires on focused environmental exposures, including those not captured in the military databases. A third laboratory approach will identify, in an exploratory study, the global DNA methylation epigenetic changes, microRNA and mRNA profiles in peripheral blood and muscle tissues from 18 subjects (six PM and six DM compared to six non-myositis controls enrolled in the second approach) and assess the effects of selected environmental exposures on these parameters. These complementary approaches should enhance the understanding of environmental factors and possible mechanisms associated with the development of myositis in the military, and provide insights into environmental risk factors that may also be relevant to the development of myositis in non-military populations.

ELIGIBILITY:
* ELIGIBILITY CRITERIA:

For Aim 1 of the study:

The inclusion criteria for myositis subjects are:

-Diagnosis of PM, DM or IBM during military service. Subjects may be active duty or no longer active duty personnel. A matrix diagnosis of myositis will be based on ICD-9 codes, laboratory tests and medical records in an attempt to match criteria for probable or definite PM, DM or IBM

The inclusion criteria for matched control subjects are:

-The same gender, race, age within 10 years, and service in the military within 10 years as the myositis subject.

The exclusion criteria for control subjects are:

-A matrix diagnosis of autoimmune or chronic muscle disease based on ICD-9 codes and medical records.

For Aims 2 and 3 of the study:

The inclusion criteria for enrollment of myositis subjects are:

* Diagnosis of myositis during military service or service as a military contractor or civilian working for the military, based on criteria for probable or definite PM or DM, or clinically or pathologically defined or possible IBM. Subjects may be active duty or no longer active duty personnel. Military contractors or civilians working for the military include those with at least 1 year of collective service on a military base or who actively deployed with military units after October 1998 and developed myositis will be eligible for this study.
* Able and willing to give informed consent, to complete the questionnaires and to donate blood samples.

The inclusion criteria for matched controls are:

* Persons with military experience or having served as a military contractor or civilian working for the military attending the same clinic or hospital as the myositis subject to which they are matched, or if not available, volunteers from the general community (such as other participating military or VA hospitals, private HCPs, or the NIH healthy volunteer program), gender- race- and age- (within 10 years) and military service period (within 10 years) matched to the myositis subject. Military contractors include those with at least 1 year of collective service on a military base or who actively deployed with military units after October 1998.
* Controls should be without a recognized autoimmune or chronic muscle disease, able and willing to give informed consent, to complete the questionnaires and to donate blood samples.

The exclusion criteria for all protocol subjects are:

* Medical illness that in the judgment of the investigators does not allow safe blood draws or other clinical evaluations needed for study participation.
* Chronic muscle diseases other than idiopathic inflammatory myopathy (e.g., infectious, dystrophic, metabolic, toxic or drug-induced myopathies).
* Cognitive impairment.
* Not able or willing to give informed consent.
* Age <18 years.
* Current incarceration

There are no gender or ethnic restrictions to enrollment in the study.

HIV is not an exclusion for this study for the two following reasons:

* It has no impact on study procedures or tests.
* HIV may be one of the viral risk factors we are investigating.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Myositis patients include diagnosis of myositis during military service or service as a military contractor based on criteria for probable or definite PM or DM, or clinically or pathologically defined or possible IBM. Subjects may be active duty or no longer active duty personnel. Military contractors include those with at least 1 year of collective service on a military base or who actively deployed with military units after October 1998 and developed myositis will be eligible for this study. Control subjects include persons with military experience or having served as a military contractor attending the same clinic or hospital as the myositis subject to which they are matched, or if not available, volunteers from the general community (such as other participating military or VA hospitals, private HCPs, or the NIH healthy volunteer program), matched to the myositis subject.
Sampling Method: Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2014-03-13 (Actual); Primary Completion 2021-10-31 (Actual)

PRIMARY OUTCOMES:
Military Myositis Questionnaire | Assessed once per respondent
  Myositis and control subjects will complete the environmnetal exposure questionnaire, a connective tissue screening questionnaire and the Patient Reported Outcomes Measurement Information System (PROMIS) Quality of Life measure to assess health related quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Adam I Schiffenbauer, M.D., Principal Investigator — National Institute of Environmental Health Sciences (NIEHS)
Locations (7):
- United States (7):
  - Miami VA Healthcare System, Miami, Florida
  - Walter Reed National Medical Center, Bethesda, Maryland
  - National Institutes of Health Clinical Center, Bethesda, Maryland
  - NIEHS Clinical Research Unit (CRU), Research Triangle Park, North Carolina
  - VA Pittsburgh Healthcare Sys., Pittsburgh, Pennsylvania
  - Naval Medical Center, Portsmouth, Portsmouth, Virginia
  - Madigan Army Medical Center, Tacoma, Washington

IPD SHARING:
Plan to Share IPD: Undecided
It is not yet known if there will be a plan to make IPD available

REFERENCES:
- [Background] Bacarese-Hamilton T, Mezzasoma L, Ardizzoni A, Bistoni F, Crisanti A. Serodiagnosis of infectious diseases with antigen microarrays. J Appl Microbiol. 2004;96(1):10-7. doi: 10.1046/j.1365-2672.2003.02111.x. PMID 14678154
- [Background] Aggarwal R, Lucas M, Fertig N, Oddis CV, Medsger TA Jr. Anti-U3 RNP autoantibodies in systemic sclerosis. Arthritis Rheum. 2009 Apr;60(4):1112-8. doi: 10.1002/art.24409. PMID 19333934
- [Background] Bach JF. The effect of infections on susceptibility to autoimmune and allergic diseases. N Engl J Med. 2002 Sep 19;347(12):911-20. doi: 10.1056/NEJMra020100. No abstract available. PMID 12239261
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2013-E-0015.html